CLINICAL TRIAL: NCT02388399
Title: Relevance of Invasively Measured Axial Plaque Stress and Wall Shear Stress Using Invasive Coronary Imaging and Hemodynamic Data
Brief Title: Invasive Measurement of Axial Plaque Stress, the Pilot Study
Acronym: REASSURE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Professor of Internal Medicine and Cardiology Deparment, Seoul National University Hospital
Other Study IDs: NCT723631
Record Dates: First submitted 2015-03-04; First posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Artery Disease
Keywords: Optical coherence tomography; Axial Plaque Stress; Wall Shear Stress; Vulnerability
MeSH Terms: conditions — Coronary Artery Disease | interventions — Equipment and Supplies; Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OCT and Pressure wire pullback tracing: This study is pilot study evaluating the feasibility of invasive measurement and estimation of hemodynamic stress acting on plaque as well as co-registration of hemodynamic data with plaque geometric data, which is obtained by optical coherence tomography
  Interventions: Procedure: Device

INTERVENTIONS:
Procedure: Device — Optical coherence tomography to evaluate plaque morphology and vulnerable features (ex> cap thickness, spotty calcification)
  Other Names: Optical coherence tomography
Procedure: Device — Resting and hyperemic pressure pullback tracing will be done with motorized pullback system.
  Other Names: Fractional flow reserve measurement with pressure pullback tracing

SUMMARY:
In this study, the investigators sought to evaluate the feasibility of estimating external hemodynamic stress acting plaque with the use of invasively measured hemodynamic data from pressure wire pullback tracing.

In addition, the investigators will also evaluate detailed plaque geometry and vulnerability using optical coherence tomography along with the hemodynamic stress.

DETAILED DESCRIPTION:
It has been well known that mechanism of acute coronary syndrome is plaque rupture and occlusion of coronary artery by this plaque rupture. Although current risk assessment for plaque rupture have mainly focused on evaluation of plaque vulnerability. However, according to the general mechanism of material failure, plaque rupture occurs whenever the external hemodynamic stress exceeds the durability of the plaque.

Recently, we evaluated the axial plaque stress, which is axial component of total traction acting on the plaque, and showed that the axial plaque stress possess significantly higher magnitude than previously known wall shear stress.

However, the axial plaque stress in our previous research was measured with computational flow dynamics analysis using coronary artery model from coronary CT angiography.

In this study, we sought to evaluate the feasibility of estimating external hemodynamic stress acting plaque with the use of invasively measured hemodynamic data from pressure wire pullback tracing.

In addition, we will also evaluate detailed plaque geometry and vulnerability using optical coherence tomography along with the hemodynamic stress.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with angina pectoris who are scheduled to do invasive coronary angiography.
* 2. Patients who have moderate (40-70%) stenosis at proximal or mid-portion of major coronary arteries.
* 3. Pressure wire pullback tracing and Optical Coherence Tomography ware successfully performed

Exclusion Criteria:

* 1. Stenosis at distal coronary or small vessel.
* 2. Patients who don't have moderate (40-70%) stenosis at proximal or mid-portion of major coronary arteries. Confirmed by invasive coronary angiography.
* 3. Inadequate quality of Optical Coherence Tomography
* 4. No data of Fractional Flow Reserve or Pressure wire pullback tracing or inadequate data of Fractional Flow Reserve or Pressure wire pullback tracing

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with angina pectoris
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Axial plaque stress (Axial component of total traction acting on the plaque) | up to 1 week
Cap thickness (measured from optical coherent tomography) | up to 1 week
  Cap thickness measured from optical coherent tomography

SECONDARY OUTCOMES:
Wall shear stress (Friction vector on the surface of the plaque) | up to 1 week
  Friction vector on the surface of the plaque
Proportion of thin cap fibrous atheroma | up to 1 week
  Plaques with cap thickness < 60um
Cardiac death and all-cause mortality | 1 year
  Between High-hemodynamic force plaque and Low-hemodynamic force plaque
Non-fatal target vessel myocardial infarction | 1 year
  Between High-hemodynamic force plaque and Low-hemodynamic force plaque
Target vessel restenosis | 1 year
  Between High-hemodynamic force plaque and Low-hemodynamic force plaque

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (4):
- South Korea (4):
  - Keimyung University Dongsan Medical Center, Daegu
  - Inje University Ilsan Paik Hospital, Goyang
  - Seoul National University Hospital, Seoul
  - Ulsan University Hospital, University of Ulsan College of Medicine, Ulsan